CLINICAL TRIAL: NCT04519320
Title: Medium and Long Term Follow-up of SARS-COV-2 Infected Patients Treated at Besançon and Dijon Hospitals: Research and Characterization of Pulmonary Sequelae
Brief Title: Medium and Long Term Follow-up of COVID-19 Infected Patients: Research and Characterization of Pulmonary Sequelae
Acronym: COV-RECUP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/499
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Respiratory Function Tests; Tomography, X-Ray Computed; Walk Test; Blood Gas Analysis; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-COV 2 Patients (Other)
  Interventions: Diagnostic Test: Pulmonary function testing

INTERVENTIONS:
Diagnostic Test: Pulmonary function testing — D0: date of first symptoms of SARS-COV-2
  M3: D0 + 3 months
  * Blood test
  * Blood gases
  * Clinical examination
  * CT Scan
  * Pulmonary function testing (PFT)
  * 6-minute walk test (6MWT)
  * MOS SF-36 Questionnaire
  * HADS scale
  * Ventilatory polygraphy
  M6: D0 + 6 months
  * Clinical examination
  * PFT
  * 6MWT
  * MOS SF-36 Questionnaire
  * HADS scale
  M12: D0 + 12 months
  * Blood test
  * Blood gases
  * Clinical examination
  * CT Scan (If anomaly found at M3)
  * PFT
  * Pulmonary Exercise Stress Test
  * 6MWT
  * MOS SF-36 Questionnaire
  * HADS scale
  Subsequent follow-up will be performed only in patients with an alteration defined by a DLCO <LLN and / or an abnormality objectified at CT-Scan attributable to SARS-CoV-2.
  M24, M36, M48 and M60: D0 + 24, 36, 48, 60 months
  * Clinical examination
  * PFT
  * 6MWT
  * MOS SF-36 Questionnaire
  * HADS scale
  Other Names: CT Scan; Six minute walk test; Pulmonary Exercise Stress Test; Blood gases; Ventilatory polygraphy; Questionnaires: HADS and MOS SF-36; Blood Test

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the cause of atypical emerging pneumonia. The clinical spectrum varies from an asymptomatic or mild illness to a serious illness with a high risk of mortality. The most severely affected patients (5%) present an acute respiratory distress syndrome (ARDS), requiring assistance with mechanical ventilation in intensive care.

In 2003, persistent lung damage was observed in a third of patients in a Singaporean cohort one year after SARS-CoV infection. A Chinese study showed that 27.3% of their SARS-CoV patients presented a decreased carbon monoxide diffusion (DLCO) and 21.5% of pulmonary fibrosis lesions.

Due to the very recent emergence of SARS-CoV-2, no data is currently available of long-term outcome of these patients. However, recent publications including short-term CT monitoring suggest the genesis of fibrotic pulmonary parenchymal sequelae.

In view of these data, the investigators can fear the occurrence of pulmonary sequelae in patients infected with SARS-CoV-2. It is therefore essential to evaluate the evolution of the respiratory status of the most severe patients who have had a stay in intensive care with respiratory assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient infected by SARS-CoV-2 (diagnosed by RT-PCR and / or typical CT imaging)
* Patient hospitalized in the intensive care units of Besançon or Dijon hospitals for severe SARS-CoV-2 pneumonia
* Postmenopausal woman for at least 24 months or surgically sterilized, or, for woman of childbearing age, use of an effective method of contraception
* Signature of informed consent to participate indicating that the subject has understood the purpose and the procedures required by the study and that he agrees to participate in the study.
* Affiliation to a French social security system .

Exclusion Criteria:

* Chronic respiratory failure under long-term oxygen therapy
* Known diffuse invasive pneumonia
* Life expectancy estimated at less than one year by the doctor
* Legal incapacity or limited legal capacity
* History of psychiatric illness, intellectual disability, lack of motivation or other conditions that may limit the understanding of informed consent
* Subject unlikely to cooperate in the study and / or weak cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant and / or lactating woman
* Subject being in the exclusion period of another study or foreseen by the "national file of the volunteers".

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with an alteration of the capillary alveolus barrier at 12 months of follow-up, characterized by a decreased of the diffusing capacity for carbon monoxide (DLCO) below the lower limit of normal | 12 months after the first symptoms of SARS-COV-2
  DLCO

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureddine S, Roux-Claude P, Laurent L, Ritter O, Dolla P, Karaer S, Claude F, Eberst G, Westeel V, Barnig C. Evaluation of long-term sequelae by cardiopulmonary exercise testing 12 months after hospitalization for severe COVID-19. BMC Pulm Med. 2023 Jan 12;23(1):13. doi: 10.1186/s12890-023-02313-x. PMID 36635717
- [Derived] Eberst G, Claude F, Laurent L, Meurisse A, Roux-Claude P, Barnig C, Vernerey D, Paget-Bailly S, Bouiller K, Chirouze C, Behr J, Grillet F, Ritter O, Karaer S, Pili-Floury S, Winiszewski H, Samain E, Decavel P, Capellier G, Westeel V. Result of one-year, prospective follow-up of intensive care unit survivors after SARS-CoV-2 pneumonia. Ann Intensive Care. 2022 Mar 9;12(1):23. doi: 10.1186/s13613-022-00997-8. PMID 35262794